CLINICAL TRIAL: NCT03761979
Title: Safety and Pharmacokinetics of Orally Administered Strontium L-Lactate in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioLink Life Sciences, Inc. (Industry)
Collaborators: Biofortis Innovation Services (Industry); NMS Laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: BIO-1703
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Low Bone Density; Osteopenia; Osteoporosis, Postmenopausal
Keywords: Bone density; Osteopenia; Osteoporosis; Bone health; Pharmacokinetics
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Intervention Model Description: This was an unblinded, sequential, three dose study. The study consisted of one screening visit (Visit 1; day -7) and three test visits (Visits 2, 3, and 4; days 0, 7, and 14) with at least a 6-d washout between test visits.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects' anonymity was maintained on electronic case report forms (eCRFs) and other documents by utilization of initials, number, or code, and not by using a subject's name. The Investigator kept a separate log showing codes, names, and addresses. All documents showing the subjects' identity were kept in strict confidence by the Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strontium dose of 170 mg (Active Comparator): The Sponsor provided each 170 mg dose of strontium as strontium L-lactate dry powder packaged in individual vials. The powder was prepared for consumption by adding 10 mL of distilled water to the vial and stirring until dissolution was complete. This liquid was then poured into an administration cup. An additional 10 mL of distilled water was used to rinse the remaining SrLac into the administration cup. Then 80 mL of distilled water was added directly into the administration cup. Following consumption of the 100 mL solution of SrLac, another 100 mL of distilled water was added into the administration cup, swirled, and consumed by the subject.
  Interventions: Dietary Supplement: Strontium L-lactate
- strontium dose of 340 mg (Active Comparator): The Sponsor provided each 340 mg dose of strontium as strontium L-lactate dry powder packaged in individual vials. The powder was prepared for consumption by adding 10 mL of distilled water to the vial and stirring until dissolution was complete. This liquid was then poured into an administration cup. An additional 10 mL of distilled water was used to rinse the remaining SrLac into the administration cup. Then 80 mL of distilled water was added directly into the administration cup. Following consumption of the 100 mL solution of SrLac, another 100 mL of distilled water was added into the administration cup, swirled, and consumed by the subject.
  Interventions: Dietary Supplement: Strontium L-lactate
- Strontium dose of 680 mg (Active Comparator): The Sponsor provided each 680 mg dose of strontium as strontium L-lactate dry powder packaged in individual vials. The powder was prepared for consumption by adding 10 mL of distilled water to the vial and stirring until dissolution was complete. This liquid was then poured into an administration cup. An additional 10 mL of distilled water was used to rinse the remaining SrLac into the administration cup. Then 80 mL of distilled water was added directly into the administration cup. Following consumption of the 100 mL solution of SrLac, another 100 mL of distilled water was added into the administration cup, swirled, and consumed by the subject.
  Interventions: Dietary Supplement: Strontium L-lactate

INTERVENTIONS:
Dietary Supplement: Strontium L-lactate — The Study Product was a highly pure form of SrLac, the strontium salt of L-lactic acid. SrLac was manufactured in compliance with current Good Manufacturing Practices. SrLac was thoroughly tested and met rigorous purity specifications. It was free from contamination by D-lactic acid and trace metals known to harm human health.
  Other Names: SrLac

SUMMARY:
No clinical trials have evaluated strontium L-lactate (SrLac), the strontium salt of the L-enantiomer of lactic acid. Therefore, this clinical study was conducted to obtain general safety and pharmacokinetic (PK) information following acute oral intakes of three doses of SrLac by healthy adults. The data provided valuable comparisons with the pharmacokinetics of other strontium salts that are in clinical use and allowed determination of the dose of SrLac that will be useful for the management of bone health.neficial for the treatment of low bone density of osteoporosis and osteopenia.

DETAILED DESCRIPTION:
Purpose: The aim of this clinical study was to obtain safety and pharmacokinetic information following acute oral intakes of three ascending doses of strontium L-lactate by healthy adults.

Subjects and methods: Ten healthy men and women, mean age 43 ± 2 years, ingested one of three ascending doses of strontium L-lactate (SrLac) once per week for three weeks in succession. Fasting blood collections were performed pre-dose and 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose for determination of serum strontium at each interval.

ELIGIBILITY:
Inclusion Criteria

1. Subject is a generally healthy male or female, 18-65 years of age, inclusive.
2. Subject has a score of 7 to l O on the Vein Access Scale at Visit l (day -7).
3. Subjects exhibits a body weight >60 kg and has a BMI of2:l 8.0 and <32.0 kg/m2 at Visit 1 (day -7).
4. Subject is willing to avoid use of any over-the-counter medications and/or dietary supplements (vitamins, minerals and/or other supplements) within 3 d prior to visit 1 (day-7) and/or prescription medications (except for stable-dose oral contraceptives) within 14 d prior to visit l (day -7) and throughout the study period.
5. Subject is willing to avoid alcohol 3 d prior to each test visit (Visits 2, 3, and 4; days 0, 7, and 14).
6. Subject is willing to avoid grapefruit and/or grapefruit juice 3 d prior to each test visit (Visits 2, 3, and 4; days 0, 7, and 14).
7. Subject is willing to maintain habitual diet, physical activity patterns, and body weight throughout the trial.
8. Subject is a non-user of all tobacco, smoking products (including, but not limited to cigarettes, cigars, chewing tobacco, e-cigarettes), and nicotine products (e.g., nicotine gum and/or nicotine patches) within 6 months of Visit 1 (day -7) and has no plans to change status during the study period.
9. Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.

l 0. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Subject has abnormal laboratory test results of clinical significance at Visit 1 (day -7) at the discretion of the Investigator. One re-test will be allowed on a separate day prior to Visit 2 (day 0), for subjects with abnormal laboratory test results.
2. Subject has a known allergy or sensitivity to any of the ingredients in the study products and/or any ingredients of the meals provided.
3. Subject has a history of anaphylaxis, a documented hypersensitivity reaction, and/or a clinically important reaction to any drug.
4. Subject has a history or presence of clinically important endocrine (including hyperparathyroidism, type l or 2 diabetes mellitus and/or hypoglycemia), cardiovascular (including, but not limited to history of myocardial infarction, peripheral arterial disease, stroke), pulmonary (including uncontrolled asthma), hepatic, renal, hematologic, immunologic, dermatologic, neurologic (such as Alzheimer's or Parkinson's patients), rheumatic (including gout), biliary, and/or psychiatric disorders (including depression and/or anxiety disorders), that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
5. Subject has had a loss of 400 mL of blood (e.g., blood/plasma donation) during the prior 30 d of visit 2 (day 0).
6. Subject has a history or current GI disorder that, in the judgment of the Investigator, may have the potential to disrupt normal digestion and absorption.
7. Subject has a history or presence of cancer in the prior two years, except for non- melanoma skin cancer.
8. Subject has a history of bariatric surgery for weight reducing purposes.
9. Subject has recently (within 6 months prior to Visit 1; day -7) had a weight loss or gain >4.5 kg.

I 0. Subject has uncontrolled hypertension (systolic blood pressure 2:160 mm Hg or diastolic blood pressure 2:100 mm Hg) as defined by the blood pressure measured at Visit 1 (day -7). One re-test will be allowed on a separate day prior to Visit 2 (day 0), for subjects with abnormal blood pressure.

11. Subject has extreme dietary habits (e.g., Atkins diet, very high protein, vegetarian, intentional consumption of a high fiber diet), in the opinion of the Clinical Investigator.

12. Subject is a female, who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.

13. Subject has been exposed to any non-registered drug product within 30 d prior to visit I (day-7).

14. Subject has a recent history of (within 12 months of screening; Visit I; day -7) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink= 12 oz beer, 5 oz wine, or I Yi oz distilled spirits).

15. Individual has a condition the Clinical Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
iAUC-0.25-12h | 0.25 hour pre-dosing to 12 hours post-dosing on each day of dosing
  The primary outcome variable was the incremental area under the curve (iAUC) for serum strontium from pre-product consumption (t = -0.25 h) to 12 h (iAUC-0.25-12h).

SECONDARY OUTCOMES:
(iAUC-0.25-∞) | 0.25 hour pre-dosing to 12 hours post-dosing on each day of dosing
  iAUC for serum strontium from pre-product consumption (t = -0.25 h) to infinity (iAUC-0.25-∞)
Cmax | 0.25 hour pre-dosing to 12 hours post-dosing on each day of dosing
  Maximum serum concentration (Cmax)
Tmax | 0.25 hour pre-dosing to 12 hours post-dosing on each day of dosing
  Time to Cmax (Tmax)
K | 0.25 hour pre-dosing to 12 hours post-dosing on each day of dosing
  Rate of elimination (K)
t1/2 | 0.25 hour pre-dosing to 12 hours post-dosing on each day of dosing
  Half life (t1/2)
Oral bioavailability (F) | 0.25 hour pre-dosing to 12 hours post-dosing on each day of dosing
  The fraction of the amount of strontium given orally that reaches the systemic circulation

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Sanoshy, Study Director — Biofortis Innovation Services
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared as needed to complete Institutional Review Board (IRB) reviews, enable statistical analyses, and prepare study reports.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3/1/2017 - 7/17/2017
Access Criteria: Access must be authorized by Study Director at Biofortis Innovation Services

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT03761979/Prot_SAP_000.pdf